CLINICAL TRIAL: NCT02628600
Title: An Open-Label Safety Extension Study to a Multicenter Study of Liposomal Amikacin for Inhalation (LAI) in Adult Patients With Nontuberculous Mycobacterial (NTM) Lung Infections Caused by Mycobacterium Avium Complex (MAC) That Are Refractory to Treatment
Brief Title: Open-label Safety Extension Study Assessing Safety and Tolerability of LAI in Patients Who Participated in Study INS-212
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS-312; 2015-003170-33 (EudraCT Number)
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: NTM Lung Infection Due to MAC
Keywords: ALIS; ARIKAYCE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prior LAI + Multidrug Regimen (Experimental): Participants in the prior Study INS-212 who received LAI+MDR. All participants in this safety extension study received LAI+MDR.
  Interventions: Drug: LAI 590 mg; Drug: Multi-drug regimen
- Prior Multidrug Regimen Alone (Experimental): Participants in the prior Study INS-212 who received MDR alone. All participants in this safety extension study received LAI+MDR.
  Interventions: Drug: LAI 590 mg; Drug: Multi-drug regimen

INTERVENTIONS:
Drug: LAI 590 mg — LAI 590 mg QD: administered by inhaling drug product that had been aerosolized in an investigational eFlow nebulizer over approximately 14 minutes
  Other Names: Amikacin Liposome Inhalation Suspension (ALIS); ARIKAYCE®
Drug: Multi-drug regimen — Multidrug antimycobacterial regimen from study INS-212

SUMMARY:
This is an open-label safety extension study to assess the safety and tolerability of once daily dosing of 590 mg Liposomal Amikacin for Inhalation (LAI) added to a multi-drug regimen in participants with nontuberculous mycobacterial (NTM) lung infections due to Mycobacterium avium complex (MAC) who were refractory to therapy and failed to convert in Study INS-212 (NCT02344004).

DETAILED DESCRIPTION:
Safety and tolerability of once daily dosing of 590 mg Liposomal Amikacin for Inhalation (LAI) added to a multi-drug regimen in participants with non-tuberculous mycobacterium (NTM) lung infections due to Mycobacterium avium complex (MAC) who are refractory to therapy and failed to convert in Study INS-212.

Participants participating in Study INS-212 who had not achieved the INS-212 protocol definition of culture conversion (3 consecutive monthly negative sputum cultures) or who had experienced a relapse or recurrence (agar positive or more than 2 consecutive broth positive results after culture conversion had occurred) by Month 6, as determined by their sputum culture results from Day 1 through Month 6 and confirmed at their scheduled Month 8 visit, were eligible to participate in Study INS-312. For participants who chose to participate in Study INS-312, the Month 8 visit of Study INS-212 became their end of treatment (EOT) visit; these participants were then asked to provide written informed consent for Study INS-312 and were enrolled directly into Study INS-312 after having met all eligibility criteria.

Participants in Study INS-212 had either received 590 mg LAI plus an MDR (LAI + MDR arm) or a multidrug regimen alone (MDR alone arm). All participants in this safety extension study were to continue the multidrug antimycobacterial regimen that they were receiving during Study INS-212 and will receive LAI 590 mg administered daily (QD) for up to 12 months. The participants will remain in the study for up to a total of 13 months (up to 12 months on-treatment plus 1 month off LAI treatment for safety follow up).

ELIGIBILITY:
Key Inclusion Criteria:

1. had successfully completed the Month 6 and End of Treatment visits in Study INS-212
2. had not achieved the INS-212 protocol definition of culture conversion by Month 6 in Study INS-212 OR had experienced a relapse or recurrence by Month 6 in Study INS-212.

Key Exclusion Criteria:

1. achieved culture conversion without relapse or recurrence in the Study INS-212 study by Month 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mange, MD, Study Director — Insmed Incorporated

REFERENCES:
- [Derived] Yamazaki Y, Nakagawa T, Jumadilova Z, Yuen D, Villa R, Hasegawa N. Management and Resolution of Hypersensitivity Pneumonitis-Related Events in Japanese Patients Treated with Amikacin Liposome Inhalation Suspension in the CONVERT and INS-312 Clinical Trials. Infect Dis Ther. 2025 Nov 4. doi: 10.1007/s40121-025-01247-7. Online ahead of print. PMID 41186908
- [Derived] Winthrop KL, Flume PA, Thomson R, Mange KC, Yuen DW, Ciesielska M, Morimoto K, Ruoss SJ, Codecasa LR, Yim JJ, Marras TK, van Ingen J, Wallace RJ Jr, Brown-Elliott BA, Coulter C, Griffith DE. Amikacin Liposome Inhalation Suspension for Mycobacterium avium Complex Lung Disease: A 12-Month Open-Label Extension Clinical Trial. Ann Am Thorac Soc. 2021 Jul;18(7):1147-1157. doi: 10.1513/AnnalsATS.202008-925OC. PMID 33326356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Study INS-212 had either received 590 mg LAI plus an MDR (LAI + MDR arm) or a multidrug regimen alone (MDR alone arm). All participants in this safety extension study, INS-312, were to continue the multidrug antimycobacterial regimen that they were receiving during Study INS-212 and received LAI 590 mg QD for up to 12 months.
Period: Overall Study
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
Started | 73 | 90
Participant Discontinued the Study | 24 | 32
Completed | 49 | 58
Not Completed | 24 | 32
Not completed — Death | 2 | 1
Not completed — Adverse Event | 3 | 20
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 2
Not completed — Other not specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population, defined as participants who received at least 1 dose of LAI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone | Total
Number analyzed (Participants) | 73 | 90 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.12) | 64.8 (10.33) | 64.8 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 105
  Male | 22 | 36 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 22 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 41 | 60 | 101
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as those AEs that occurred on or after the date of first dose of study medication in INS-312 and within 28 days after the last dose. If it couldn't be determined whether the AE is treatment emergent due to a partial onset date, then it was classified as treatment emergent.
Time Frame: From baseline to 28 days after end of treatment, up to 13 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
Number analyzed (Participants) | 73 | 90
participants
  ≥1 Treatment-emergent AE (TEAE) | 68 | 90
  ≥1 Serious TEAE (sTEAE) | 20 | 32
  ≥1 TEAE leading to study drug withdrawn | 8 | 24
  ≥1 TE AE Leading to LAI withdrawn | 6 | 22
  ≥1 TEAE Leading to MDR for NTM withdrawn | 4 | 8
  ≥1 TEAE Leading to LAI and MDR for NTM withdrawn | 1 | 5
  ≥1 sTEAE leading to LAI withdrawn | 3 | 9
  ≥1 TEAE leading to death | 2 | 4

2. Secondary Outcome: Number of Participants Achieving Culture Conversion by Month 6 and Month 12
Description: 6 months: Converters are defined as participants who had 3 consecutive monthly MAC-negative sputum cultures by Month 6 (last opportunity to convert was at Month 4).
  12 months: Converters are defined as participants who had 3 consecutive monthly MAC-negative sputum cultures by Month 12 (last opportunity to convert was at Month 10).
Time Frame: by Month 6 and Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
Number analyzed (Participants) | 73 | 90
Participants
  6 months | 7 | 24
  12 months | 10 | 30

3. Secondary Outcome: Time to Culture Conversion
Description: The time to culture conversion is defined as the date of conversion for participants achieving culture conversion is defined as the date of the first of 3-consecutive monthly negative sputum cultures. Then, the number of days to culture conversion is defined as the difference between the date of conversion and the date of first dose of LAI.
Time Frame: by Month 12
Population: The Safety population was the set of all enrolled participants who received at least 1 dose of LAI.
Measure: Median (Full Range); unit: months
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
Number analyzed (Participants) | 73 | 90
months | NA [NA to NA] — Not able to be estimated due to an insufficient number of participants achieving conversion | NA [NA to NA] — Not able to be estimated due to an insufficient number of participants achieving conversion

4. Secondary Outcome: Change From Baseline (Day 1) to Month 6 and Month 12 in the 6MWT Distance
Description: A 6-minute walk assessment of exertional capability was performed at Baseline (Day 1) and Month 6 and Month 12/EOT. The standardized protocol based on the American Thoracic Society (ATS) guidelines (http://doi.org/10.1164/ajrccm.166.1.at1102) was used. After assessments were performed for heart rate, blood pressure, pulse oximetry (SpO2), dyspnea, and overall fatigue using the Borg scale, participants were instructed to walk on a prescribed course as far as they could in 6 minutes. Pre-test assessment parameters were repeated after exertion. The maximum distance achieved and post exertion heart rate and SpO2 were compared to pre-test values. The maximum distance achieved was recorded in the electronic case report form.
Time Frame: From baseline to Month 12 or end of treatment
Population: Baseline: number of participants with data at this visit.
  Change from baseline: number of participants with both baseline and 6 month scores.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
Number analyzed (Participants) | 73 | 90
meters
  Baseline: number analyzed (Participants) | 58 | 71
  Baseline | 435.9 (132.33) | 449.0 (122.64)
  Change from Baseline to Month 6: number analyzed (Participants) | 58 | 71
  Change from Baseline to Month 6 | -10.4 (69.77) | -20.8 (51.57)
  Change from Baseline to Month 12: number analyzed (Participants) | 47 | 56
  Change from Baseline to Month 12 | -10.1 (79.23) | -42.2 (72.66)

ADVERSE EVENTS:
Time Frame: From baseline up to 28 days after end of treatment, up to 13 months
Arm/Group | Prior LAI + Multidrug Regimen | Prior Multidrug Regimen Alone
All-Cause Mortality (participants affected / at risk) | 2/73 | 4/90
Serious Adverse Events (participants affected / at risk) | 20/73 | 32/90
Other Adverse Events (participants affected / at risk) | 45/73 | 75/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior LAI + Multidrug Regimen (N=73) | Prior Multidrug Regimen Alone (N=90)
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cataract (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 3
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 2 | 5
Pneumonia (Infections and infestations) | 3 | 4
Pneumonia fungal (Infections and infestations) | 0 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinobronchitis (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior LAI + Multidrug Regimen (N=73) | Prior Multidrug Regimen Alone (N=90)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 9 (11)
Nausea (Gastrointestinal disorders) | 5 (6) | 9 (10)
Fatigue (General disorders) | 3 (3) | 13 (13)
Nasopharyngitis (Infections and infestations) | 10 (11) | 7 (10)
Infective exacerbation of bronchiectasis (Infections and infestations) | 6 (7) | 10 (10)
Weight decreased (Investigations) | 7 (7) | 8 (8)
Haematuria (Renal and urinary disorders) | 4 (4) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 39 (54)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 32 (37)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 16 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees not to originate or use the name of Insmed Incorporated, or study drug code in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment to the protocol, or to the performance of this protocol, without the prior written consent of Insmed Incorporated.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT02628600/SAP_000.pdf
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02628600/Prot_001.pdf